CLINICAL TRIAL: NCT03144908
Title: Medical Provider Experience and Assessment on Healthcare Decisions Regarding Dietary and Environmental Allergen Exposure
Brief Title: Healthcare Decisions on Dietary and Environmental Allergen Exposure
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Data Collection Analysis Business Management (Other)
Collaborators: PAS Research Services (Other)
Responsible Party: Sponsor
Other Study IDs: PAS1462
Record Dates: First submitted 2017-05-02; First posted 2017-05-09 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Dietary Allergy; Environmental Allergy
MeSH Terms: conditions — Environmental Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard Operating Procedures — Observational on Standard Operating Procedures

SUMMARY:
Design of this study is to collect data and review Principal Investigators standard operating procedures on allergy testing and changes made to their specific SOP.

DETAILED DESCRIPTION:
The purpose of this minimal risk observational study is to increase surveillance for dietary and environmental allergens exposure and to also determine targeted risk reducing and preventative strategies.

ELIGIBILITY:
Inclusion Criteria:

* Must be a medical practitioner Medical Doctor (MD) Doctor of Osteopathic (DO) Physician Assistant (PA) Advanced Practice Registered Nurse (APRN) Nurse Practioner (NP) Must have a current standard operating procedure that includes obtaining/reviewing medical history and family medical history.

Exclusion Criteria:

* Government funded insurance data cannot be included in the study

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Only licensed providers, as per the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Provider Structures and Processes | 36 months
  Plan of Care Changes due to Allergy testing. Provider based observational survey system on the health and well being of patients and populations.

CONTACTS AND LOCATIONS:
Locations (1):
- DCABM, Land O' Lakes, Florida, United States